CLINICAL TRIAL: NCT06626633
Title: Phase 1 Clinical Trial of the STING Agonist CRD3874-SI in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: 2321GCCC: CRD3874-SI in Patients With Relapsed/Refractory AML
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2321GCCC ; HP-00105008
Record Dates: First submitted 2024-08-01; First posted 2024-10-04 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: STING agonist CRD3874-SI in patients with relapsed/refractory acute myeloid leukemia
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- STING agonist CRD3874-SI in patients with relapsed/refractory acute myeloid leukemia (Experimental): Drug Product: CRD3874 solution for injection (CRD3874-SI) Type of drug: Synthetic small molecule Formulation: Sterile solution of CRD3874 for injection Route of Administration: IV infusion over one hour Strength: 6 mg/mL Schedule: Cycle: once weekly infusion x 4 (Days 1, 8, 15 and 22) over 28-day for Cycles 1 and 2. For Cycle 3 and onward, weekly infusion x 3 (Days 1, 8 and 15), until they develop unacceptable toxicities or disease progression, or do not achieve at least a morphologic leukemia-free state response after 6 cycles.
  Interventions: Drug: CRD3874

INTERVENTIONS:
Drug: CRD3874 — CRD3874-SI is a STING agonist. CRD3874 is a synthetic drug that activates STING, and STING stimulates the immune system to kill cancer cells. In experiments on blood from humans, CRD3874 makes blood cells produce molecules responsible for anti-cancer activity. CRD3874 was tested in mice with cancers including leukemia, head and neck cancer, lung cancer, pancreatic cancer and sarcoma. In these mice, CRD3874 made tumors shrink or disappear, and some mice developed long-lasting immunity against cancer.

SUMMARY:
This clinical research study is being done to answer questions about how to treat cancer.

To clear cancer cells from the body, the immune system needs the action of proteins called Type 1 interferons. The protein STING (for STimulator of INterferon Genes) stimulates the body to make Type 1 interferons. Type 1 interferons activate key molecules in cancer immunity to kill cancer cells.

CRD3874 is a synthetic drug that activates STING, and STING stimulates the immune system to kill cancer cells. In experiments on blood from humans, CRD3874 makes blood cells produce molecules responsible for anti-cancer activity. CRD3874 was tested in mice with cancers including leukemia, head and neck cancer, lung cancer, pancreatic cancer and sarcoma. In these mice, CRD3874 made tumors shrink or disappear, and some mice developed long-lasting immunity against cancer. Also, when CRD3874 was given with other anti-cancer treatments, it increased their anti-cancer effects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age ≥ 18 years at the time of signing the ICF
* Able to understand and willing to provide written informed consent
* Willing to comply with clinical study instructions and requirements.
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2 (Appendix 1).
* Pathologically confirmed diagnosis of AML by 2022 International Consensus Classification of Myeloid Neoplasms and Acute Leukemias criteria (2)
* AML may be de novo, following a prior hematologic disorder including myelodysplastic syndrome or Philadelphia chromosome-negative myeloproliferative neoplasm, and/or therapy-related
* Patients must have relapsed/refractory AML, with any prior therapies and any number of prior therapies, and have no further standard therapies available.
* Any prior therapy must have been completed ≥2 weeks prior to Day 1 of treatment on study, and all treatment-related adverse events (except alopecia) should have recovered to <Grade 1.
* Hematologic abnormalities that are thought to be primarily related to leukemia are not considered to be toxicities and do not need to resolve to <Grade 1.
* Myeloid growth factors must have been stopped ≥1 week (filgrastim) or ≥2 weeks (pegfilgrastim) before starting study treatment.
* Prior autologous hematopoietic stem cell transplantation is allowed.
* Prior allogeneic hematopoietic stem cell transplantation is also allowed, if patients are ≥60 days from stem cell infusion, have no evidence of graft-versus-host disease (GVHD) >Grade 1, and are >4 weeks off calcineurin therapy and ≥2 weeks off all immunosuppressive therapy.
* Peripheral blast count must be <50 × 109/L. Hydroxyurea is permitted for blast count control before starting study treatment, but must be stopped ≥24 hours before starting study treatment. It may be reintroduced per physician decision if >50 × 109/L blasts recur during treatment Cycle 1 and managed per physician decision.
* Patients with other malignancies are allowed, if other malignancies are inactive and not requiring concurrent therapy except hormonal therapy for stable breast or prostate cancer.
* Aspartate aminotransferase (AST) must be <2.5 x Upper Limit Normal (ULN), alanine aminotransferase (ALT) <2.5 x ULN and total serum bilirubin <1.5 x ULN unless thought due to hemolysis or Gilbert's Syndrome.
* Adequate renal function as defined by calculated creatinine clearance (CrCl) >60 ml/minute by the Cockcroft-Gault formula
* Left ventricular ejection fraction (LVEF) >50%, as measured by echocardiogram (2D-ECHO)
* Life expectancy of at least three months at screening, according to the Investigator's opinion
* Women of childbearing potential (defined as a sexually mature female who has not undergone a hysterectomy or bilateral oophorectomy or who has not been naturally postmenopausal for at least 24 consecutive months) must have a negative serum or urine pregnancy test within 7 days of study entry.
* Women of childbearing potential and sexually active men with female partners of childbearing potential must agree to use effective contraception, including abstinence or two forms of contraception, during study treatment and for four weeks after the last dose odf study drug.

Exclusion Criteria:

* Acute promyelocytic leukemia
* Blast phase of chronic myeloid leukemia
* Known active central nervous system leukemia
* Concurrent chemotherapy, radiation therapy, immunotherapy or other investigational agents
* Active, uncontrolled infection
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements in the investigator's judgment
* Malignancies other than AML requiring active therapy except hormonal therapy for stable breast or prostate cancer
* Active autoimmune disease other than vitiligo, type 1 diabetes, or controlled hypothyroidism
* Interstitial lung disease or any disease requiring supplemental oxygen, or history of pneumonitis or pulmonary fibrosis from any cause
* Known prior severe hypersensitivity to an investigational product or any component of the study drug therapy's formulations including polyethylene glycol (PEG; National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] v5.0 Grade ≥ 3)
* Prior chemotherapy or targeted small molecule therapy within 3 weeks, anticancer monoclonal antibody within four weeks or five half-lives, if shorter, or radiation therapy within 2 weeks prior to the first CRD3874-SI infusion prior to study Day 1, or not recovered (i.e., Grade ≤ 1 or at baseline) from AE due to a previously administered agent (Note: Alopecia is acceptable. If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study therapy)
* Prior organ transplantation, other than allogeneic or autologous hematopoietic stem cell transplantation.
* Currently participating in a study and receiving study therapy, or participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment or 5 half-lives, whichever is longer.
* Received a live vaccine within 30 days of the planned start of study drug. (Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines and are not allowed.)
* Evidence of clinically significant immunosuppression including the following:

  * Primary immunodeficiency state such as SCID
  * Concurrent opportunistic infection
* Receiving systemic immunosuppressive therapy (>2 weeks) including oral steroid doses > 10 mg/day of prednisone or equivalent within seven days prior to enrollment. In the setting of non-immune mediated indications for use, chronic/active low dose steroid use (equivalent to ≤ 10 mg/day prednisone) may be permitted at the discretion of the Principal Investigator (Note: Other steroid formulations or steroid use for other indications may be permitted and include: 1) Intranasal, inhaled, ocular, or topical steroids, or local steroid injection (e.g., intra-articular injection); 2) Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; 3) Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* History or evidence of symptomatic autoimmune disease (e.g., pneumonitis, glomerulonephritis, vasculitis, or other), or history of active autoimmune disease that has required systemic treatment (i.e., use of corticosteroids, immunosuppressive drugs or biological agents used for treatment of autoimmune diseases) in past two years prior to enrollment (Note: Replacement therapy [e.g., thyroxine for hypothyroidism, insulin for diabetes or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency] is not considered a form of systemic treatment for autoimmune disease.)
* Evidence of clinically significant interstitial lung disease, history of interstitial lung disease, or active, noninfectious pneumonitis related to prior immunotherapy treatment
* Uncontrolled medical condition including current active infection requiring systemic therapy or symptomatic congestive heart failure (CHF) within six months that in the Investigator's opinion compromises the ability of the participant to complete all study-related requirements safely
* Mean resting corrected QTcF interval ≥ 470 ms on a 12-lead electrocardiogram (ECG) for males and females
* History of unstable or deteriorating cardiovascular disease within the previous six months prior to screening, including but not limited to the following:

  * Unstable angina or myocardial infarction (MI)
  * Cerebrovascular accident (CVA)/stroke
  * CHF (New York Heart Association [NYHA] Class III or IV)
  * Uncontrolled clinically significant arrhythmias
* Known to be positive for active Hepatitis B (HBV; Hepatitis B surface antigen [HBsAg] reactive with detectable HBV DNA), or Hepatitis C (HCV; detectable HCV RNA [qualitative])

  * Patients with chronic HBV (positive HBsAg and/or Hepatitis B core antibody [HBcAb] and negative HBV DNA by polymerase chain reaction [PCR]) are eligible for this study if they are on suppressive antiviral therapy and deemed safe by a gastroenterologist
  * Patients who are HCV antibody (Ab)-positive but HCV RNA-negative due to prior treatment or natural resolution will be considered eligible
* Known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies) disease that is not controlled. Individuals known to be HIV-positive will be considered eligible if all the following criteria are met:

  * Established antiretroviral treatment (ART) for at least four weeks and have an HIV viral load less than 400 copies/mL prior to enrollment
  * CD4+ T-cell counts ≥ 350 cells/uL
  * No opportunistic infection within the past 12 months
* No known history of active tuberculosis (TB)
* The presence of a concurrent active malignancy that in the opinion of the Investigator could compromise the conduct of the study or interfere with determining the outcomes of the study objectives
* Women who are pregnant or breastfeeding
* Expecting to conceive or father children within the projected duration of the study, starting with the prescreening or screening visit through three months after the last dose of study treatment(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2024-08-26 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability by multiplex cytokine profiling | 2 years
  To evaluate the safety and tolerability of CRD3874-SI (a STING agonist) in patients with relapsed/refractory acute myeloid leukemia and to determine the biologically effective dose and recommended Phase 2 dose (RP2D).
  Exploratory studies will include measurement of additional cytokines including IFNα, IL-1α, IL-1β, IL-10, IFN-γ, TNFα, MCP-1 and GM-CSF by multiplex cytokine profiling
Safety and Tolerability by qPCR | 2 years
  To evaluate the safety and tolerability of CRD3874-SI (a STING agonist) in patients with relapsed/refractory acute myeloid leukemia and to determine the biologically effective dose and recommended Phase 2 dose (RP2D).
  STING and immediate downstream targets (IRF3, IRF7, TBK1, STAT6) and NFKB pathway (GADD45a, TNFx, JUNB, NFKB2, IL7R, IKK) and IFN pathway (IFNB, ISG15, ISG20, IFI27, IFI44) targets by qPCR,
Safety and Tolerability by Western blot analysis | 2 years
  To evaluate the safety and tolerability of CRD3874-SI (a STING agonist) in patients with relapsed/refractory acute myeloid leukemia and to determine the biologically effective dose and recommended Phase 2 dose (RP2D).
  STING and downstream targets including TBK1, IRF3 and IRF7, STAT6 and TNFx and phosphorylated/activated counterparts by Western blot analysis
Safety and Tolerability by colony formation assays | 2 years
  To evaluate the safety and tolerability of CRD3874-SI (a STING agonist) in patients with relapsed/refractory acute myeloid leukemia and to determine the biologically effective dose and recommended Phase 2 dose (RP2D).
  Bcl-2 family proteins by Western blot analysis, apoptosis by flow cytometry and clonogenic potential by colony formation assays.

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | 2 years
  PK parameters will include area under the curve (AUC) in ng·hr/mL
Peak Plasma Concentration (Cmax) | 2 years
  PK parameters will include maximum concentration (Cmax) in ng/mL
Trough Concentration (Ctrough) | 2 years
  PK parameters will include trough concentration (Ctrough) in ng/mL. Blood samples will be collected. Plasma will be used for PK studies.
Pharmacodynamic (PD) effects of CRD3874-SI | 2 years
  PD endpoint will be measurement of STING pathway-relevant cytokines CXCL10, IL6 and IFNβ levels in plasma.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States